CLINICAL TRIAL: NCT06681441
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, 3-way Cross-over Study to Assess the Pharmacodynamic Effects of Two-dose Levels of QRL-101 on Transcranial Magnetic Stimulation and Nerve Excitability Threshold Tracking in Healthy Participants
Brief Title: A 3-way Cross-over Study on the Effects of QRL-101 on Transcranial Magnetic Stimulation and Nerve Excitability in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QurAlis Corporation (Industry)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: QRL-101-05
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: QRL-101

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, 3-way cross-over, single-dose study to investigate the effects of QRL-101 on TMS-EMG-EEG, mNETT, and pEEG in healthy participants.
Who Masked: Participant, Investigator
Masking Description: A participant and investigator-blinded, randomized, placebo-controlled design will be used to minimize bias in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Group 1 (Experimental): Participants will be randomized into 1 of 6 treatment sequences in a 3-way cross-over
  Interventions: Drug: QRL-101 Dose A; Drug: QRL-101 Dose B; Drug: Placebo
- Treatment Group 2 (Experimental): Participants will be randomized into 1 of 6 treatment sequences in a 3-way cross-over
  Interventions: Drug: QRL-101 Dose A; Drug: QRL-101 Dose B; Drug: Placebo
- Treatment Group 3 (Experimental): Participants will be randomized into 1 of 6 treatment sequences in a 3-way cross-over
  Interventions: Drug: QRL-101 Dose A; Drug: QRL-101 Dose B; Drug: Placebo
- Treatment Group 4 (Experimental): Participants will be randomized into 1 of 6 treatment sequences in a 3-way cross-over
  Interventions: Drug: QRL-101 Dose A; Drug: QRL-101 Dose B; Drug: Placebo
- Treatment Group 5 (Experimental): Participants will be randomized into 1 of 6 treatment sequences in a 3-way cross-over
  Interventions: Drug: QRL-101 Dose A; Drug: QRL-101 Dose B; Drug: Placebo
- Treatment Group 6 (Experimental): Participants will be randomized into 1 of 6 treatment sequences in a 3-way cross-over
  Interventions: Drug: QRL-101 Dose A; Drug: QRL-101 Dose B; Drug: Placebo

INTERVENTIONS:
Drug: QRL-101 Dose A — All participants will receive three single-dose oral administrations in randomized order, scheduled across three separate study visits, with a 7-day washout period between each visit.
Drug: QRL-101 Dose B — All participants will receive three single-dose oral administrations in randomized order, scheduled across three separate study visits, with a 7-day washout period between each visit.
Drug: Placebo — All participants will receive three single-dose oral administrations in randomized order, scheduled across three separate study visits, with a 7-day washout period between each visit.

SUMMARY:
This is a phase I, prospective, single-center, randomized, double-blind, placebo-controlled, three-way cross-over study to evaluate the safety and tolerability of QRL-101 and investigate the pharmacodynamic effects of two dose levels of QRL-101 on transcranial magnetic stimulation (TMS) and nerve excitability threshold tracking (NETT) in healthy participants.

After screening and training, participants will be randomized to one of six treatment sequences of William's square balanced for first-order carry-over design consisting of two doses of QRL-101 or placebo, with at least seven days between each treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and postmenopausal women between the ages ≥ 18 and ≤ 55.
2. BMI ≥ 18.0 and ≤ 32.0 kg/m2, and body weight ≥ 50 kg, at screening.
3. Willing and able to practice effective contraception from the screening through at least 2 days after their last dose of study treatment.
4. Participants must be able to communicate effectively (in Dutch) with the study personnel and be willing to comply with the requirements of the study.

Exclusion Criteria:

1. Evidence of any acute or chronic disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study.
2. History or presence of conditions which, in the judgment of the investigator, are known to interfere with drug absorption, distribution, metabolism, or excretion.
3. History or presence of conditions which might increase the risk of performing TMS (e.g., epilepsy, febrile seizures, intracranial mass lesion, hydrocephalus, clinically significant head injury or trauma, metal objects in the brain or skull, cochlear implant or a deep brain stimulation device)
4. Any condition that could interfere with the quality of, or ability to perform, TMS (e.g., an abnormal sleeping pattern, unremovable dreadlocks or hairpieces, or a resting motor threshold (rMT) of more than 75%.

*Other inclusion and exclusion criteria may apply*

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Single pulse TMS-EMG motor evoked potential (MEP) amplitude (μV) compared to placebo | 3 study periods, with a washout period of at least 7 days between each visit. Each study period consists of 2 nights and 1 study day.
  To compare two dose levels of QRL-101 versus placebo on cortical excitability
mNETT strength-duration time constant (SDTC) compared to placebo SDTC | 3 study periods, with a washout period of at least 7 days between each visit. Each study period consists of 2 nights and 1 study day.
  To compare two dose levels of QRL-101 versus placebo on peripheral motor nerve excitability

SECONDARY OUTCOMES:
Other Single pulse TMS-EMG MEP parameters | 3 study periods, with a washout period of at least 7 days between each visit. Each study period consists of 2 nights and 1 study day.
  To compare two dose levels of QRL-101 versus placebo on cortical excitability
pEEG: power in the alpha frequency bands in resting state with eyes open and closed | 3 study periods, with a washout period of at least 7 days between each visit. Each study period consists of 2 nights and 1 study day.
  To compare two dose levels of QRL-101 versus placebo on spontaneous brain activity measured by resting state pharmaco-encephalography (pEEG)
Incidence of AEs and SAEs | 3 study periods, with a washout period of at least 7 days between each visit. Each study period consists of 2 nights and 1 study day.
  Absolute values and changes from baseline values in vital signs, clinical laboratory tests, and ECG parameters
Plasma QRL-101 concentrations | 3 study periods, with a washout period of at least 7 days between each visit. Each study period consists of 2 nights and 1 study day.
  AUC0-24

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kremer, PharmD, MD, PhD, Principal Investigator — Centre for Human Drug Research; K. (Kaye) de Cuba,, MD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands